CLINICAL TRIAL: NCT01020877
Title: A Study to Evaluate the Relative Bioavailability of Two Metronidazole Vaginal Gel Formulations
Brief Title: Bioavailability of Metronidazole Vaginal Gel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10136019
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2010-03-23 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects; Healthy, Normal Subjects
MeSH Terms: interventions — Metronidazole; Benchmarking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Metronidazole Vaginal Gel
  Interventions: Drug: Metronidazole
- 2 (Active Comparator): MetroGel-Vaginal®
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Vaginal Gel, 0.75%
  Arms: 1
Drug: Metronidazole — Vaginal Gel, 0.75%
  Other Names: MetroGel-Vaginal®
  Arms: 2

SUMMARY:
The primary object of this study was to evaluate the relative bioavailability of the test formulation of metronidazole vaginal gel with the already marketed reference formulation MetroGel-Vaginal Gel® in healthy adult female subjects.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Females, 18 years of age or older.
* Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
* Signed informed consent form, which meets all criteria of current FDA regulations.
* If female and of child bearing potential prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g. condom, IUD, oral or implanted hormonal contraceptives).
* Weight within + 25% from normal for height and weight for body frame as described in Novum Standard Operating Procedures adapted from the "MetLife® Height and Weight Tablets", Copyright© 1993.

Exclusion Criteria:

* Females who are pregnant, lactating, or likely to become pregnant during the study.
* History of allergy or sensitivity to metronidazole, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* Significant history or current evidence of chronic infectious disease, system disorder or organ disorder.
* History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
* Presence of a medical condition requiring regular treatment with prescription drugs (other than contraceptives or hormonal replacement therapy).
* Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
* Receipt of any drug as part of a research study within 30 days prior to dosing.
* Drug or alcohol addiction requiring treatment in the past 12 months.
* Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days prior to dosing.
* Positive test for HIV, Hepatitis B surface antigen or Hepatitis C antibody.
* Positive test results for drugs of abuse at screening.
* Evidence of vulvovaginitis or cervicitis (e.g. Bacterial vaginosis, vaginal candidiasis, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhea, or history of Herpes simplex or human papillomavirus).
* Vulvar or vaginal conditions that may affect absorption of the drug.
* Clinically significant abnormal findings on PAP smear within previous 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2001-11; Primary Completion 2001-11 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley A Kennedy, MD, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Metronidazole) First: 0.75% Metronidazole Vaginal Gel test product dosed in first period followed by 0.75% MetroGel-Vaginal® reference product dosed in the second period.
- Reference (MetroGel-Vaginal®) First: 0.75% MetroGel-Vaginal® reference product dosed in first period followed by 0.75% Metronidazole Vaginal Gel test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Metronidazole) First | Reference (MetroGel-Vaginal®) First
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Test (Metronidazole) First | Reference (MetroGel-Vaginal®) First
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test (Metronidazole) First | Reference (MetroGel-Vaginal®) First
Started | 19 | 19
Completed | 18 | 19
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Metronidazole) First | Reference (MetroGel-Vaginal®) First | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 4 | 8 | 12
  Caucasian | 13 | 11 | 24
  More Than One | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed. One subject had very low plasma metronidazole levels for Period I samples, therefore the data from this subject was dropped from the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Metronidazole): 0.75% Metronidazole Vaginal Gel test product dosed in either period.
- Reference (MetroGel-Vaginal®): 0.75% MetroGel-Vaginal® reference product dosed in either period.
Arm/Group | Test (Metronidazole) | Reference (MetroGel-Vaginal®)
Number analyzed (Participants) | 36 | 36
ng/mL | 281.111 (72.222) | 257.194 (71.228)
Statistical Analysis 1: Comparison: Test (Metronidazole) vs Reference (MetroGel-Vaginal®); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test[T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 110, 90% CI 2-sided [103 to 117] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 60 hour period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Metronidazole) | Reference (MetroGel-Vaginal®)
Number analyzed (Participants) | 36 | 36
ng*h/mL | 5921.046 (1713.316) | 5593.855 (1683.155)
Statistical Analysis 1: Comparison: Test (Metronidazole) vs Reference (MetroGel-Vaginal®); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 106, 90% CI 2-sided [98.2 to 115] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 60 hour period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Metronidazole) | Reference (MetroGel-Vaginal®)
Number analyzed (Participants) | 36 | 36
ng*h/mL | 5989.237 (1737.791) | 5693.259 (1735.116)
Statistical Analysis 1: Comparison: Test (Metronidazole) vs Reference (MetroGel-Vaginal®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of the T/R geometric mean x 100 = 106, 90% CI 2-sided [97.6 to 115] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 2 weeks in duration
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Test (Metronidazole) | Reference (MetroGel-Vaginal®)
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 10/38 | 16/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Metronidazole) (N=38) | Reference (MetroGel-Vaginal®) (N=38)
Headache (General disorders) | 6 (7) | 8 (9)
Nausea (General disorders) | 1 (1) | 2 (3)
Blood in Urine (General disorders) | 1 (1) | 2 (2)
Diarrhea (General disorders) | 0 (0) | 2 (2)
Abdominal Pain/Cramps (General disorders) | 2 (2) | 0 (0)
Protein in Urine (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.